CLINICAL TRIAL: NCT00756249
Title: Randomised, Double-blind, Placebo-controlled, Single-dose, Dose-escalation Study of the Safety, Tolerability, and Pharmacokinetics of Lu AA24493 in Acute Ischemic Stroke
Brief Title: Safety Study of Carbamylated Erythropoietin (CEPO) to Treat Patients With Acute Ischemic Stroke
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: H. Lundbeck A/S, H. Lundbeck A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11767A; 2006-005959-15 (EudraCT Number)
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2010-09-27 (Estimated); Status verified 2010-09

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Erythropoietin; Carbamylated; Neuroprotection
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Lu AA24493 (CEPO): 0.005 mcg/kg (Experimental)
  Interventions: Drug: Lu AA24493 (CEPO)
- Lu AA24493 (CEPO): 0.05 mcg/kg (Experimental)
  Interventions: Drug: Lu AA24493 (CEPO)
- Lu AA24493 (CEPO): 0.5 mcg/kg (Experimental)
  Interventions: Drug: Lu AA24493 (CEPO)
- Lu AA24493 (CEPO): 5.0 mcg/kg (Experimental)
  Interventions: Drug: Lu AA24493 (CEPO)
- Lu AA24493 (CEPO): 50.0 mcg/kg (Experimental)
  Interventions: Drug: Lu AA24493 (CEPO)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lu AA24493 (CEPO) — 0.005 - 50.0 mcg/kg body weight, IV, within 12-48 hrs from symptom onset
  Arms: Lu AA24493 (CEPO): 0.005 mcg/kg; Lu AA24493 (CEPO): 0.05 mcg/kg; Lu AA24493 (CEPO): 0.5 mcg/kg; Lu AA24493 (CEPO): 5.0 mcg/kg; Lu AA24493 (CEPO): 50.0 mcg/kg
Drug: Placebo — Vials with solution for IV infusion
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to determine whether carbamylated erythropoietin (CEPO) is a safe treatment for patients who have suffered an acute ischemic stroke.

DETAILED DESCRIPTION:
Acute ischemic stroke is a major cause of death and severe disability. There is only one approved pharmacological treatment, Alteplase, which has to be administered within 3 hours from symptom onset. Consequently, only about 2-3% of patients world wide with ischemic strokes are treated. The naturally occurring hormone, erythropoietin (EPO), is able to protect various neuronal tissues from ischemic injury and is beneficial in animal models of acute ischemic stroke. However, treatment of stroke with EPO is undesirable due to its ability to stimulate production of red blood cells and to promote the blood to coagulate. Lu AA24493 is a modified (carbamylated) version of EPO, neuroprotective but without the haematopoietic side effects. Lu AA24493 is developed for treatment of patients with acute ischemic stroke.

In this safety study of single doses with Lu AA24493, patients will receive Lu AA24493 within 12-48 hours from symptom onset.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 90 years
* Clinical diagnosis of acute ischemic stroke
* Measurable stroke-related deficit
* Patient is stable
* Treatment can be initiated between 12 hours and 48 hours after the onset of stroke
* Expected hospital stay of at least 72 hours after study medication
* If female then not of childbearing potential

Exclusion Criteria:

* Primary intracerebral haemorrhage (ICH), or parenchymal haemorrhagic transformation of infarction (type PHI or PHII as defined in ECASS), subarachnoid haemorrhage (SAH), arterio-venous malformation (AVM), cerebral aneurysm, or cerebral neoplasm
* Treated with a thrombolytic <24 hours (if >24 hours excluded ICH then eligible)
* Score >0 on the NIHSS item 1a
* Pre-stroke mRS score >1
* Uncontrolled hypertension
* Previous treatment with erythropoietin
* Clinically significant abnormal ECG
* Cerebral pathology
* Received or donated blood within previous 3 months

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) and the modified Rankin Scale (mRS) | Baseline, Day 7, Day 30; for NIHSS also Day 2 and 3

SECONDARY OUTCOMES:
Pharmacokinetics, immunogenicity and mechanistic biomarkers (S-100b, glial fibrillary acidic protein (GFAP), matrix metalloproteinase 9 (MMP-9)) | Baseline, Day 1-4, Day 7 and Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (5):
- FI004, Helsinki, Finland
- FR002, Paris, France
- NL005, Breda, Netherlands
- SG003, Singapore, Singapore
- GB001, Glasgow, United Kingdom